CLINICAL TRIAL: NCT04086407
Title: The Effect of Head Pitch and Roll Rotation Independent of Torso Rotation on the AHI in Positional Obstructive Sleep Apnea
Brief Title: Apnea Hypopnea Index Severity Versus Head Position During Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sleep Systems (Industry)
Collaborators: New England IRB (Unknown); Mass Lung and Allergy, PC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Apnea Guard - 1400
Record Dates: First submitted 2019-08-29; First posted 2019-09-11 (Actual); Results first posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Sleep Disordered Breathing; Sleep Hypopnea; Sleep Apnea; Sleep Apnea, Obstructive; Snoring
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Masking Description: Subject data is randomized to Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Forehead sensor recording precision head pitch and roll angle (Experimental): During an overnight polysomnography, participants were coached by sleep research technologists to sleep with their head in positions hypothesized to minimize apnea severity ≤20⁰ or ≥160⁰, and those hypothesized to maximize apnea severity between 30⁰ and 150⁰. Head roll angles were measured and recorded by the participant's forehead sensor attached with adhesive and tape. Extreme head positions were attempted with the torso in both supine and non-supine positions so show insensitivity to torso position. A custom interface was developed to maintain compatibility with specific bedside polysomnography recorder auxiliary inputs. Sleep epochs were considered those where the subject slept for at least 10 minutes. Each head position epoch was analyzed for apnea hypopnea index and oxygen desaturation.
  Interventions: Device: Dual-axis inclinometer attached to the subject's forehead with tape

INTERVENTIONS:
Device: Dual-axis inclinometer attached to the subject's forehead with tape — This is the first clinical trial in the industry to address OSA symptom severity and snoring as a direct function of head pitch and roll angle. The head pitch and roll angle can be used with high consistency to predict OSA symptom severity. The apnea equation is based on the gravitational crush forces of the mass of the tongue and nearby tissue on the upper air way and is valid for most OSA sufferers.

SUMMARY:
This study evaluates the correlation of the position of the head during sleep, independent of the position of the torso, and the severity of apnea hypopneas in obstructive sleep apnea.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a common diagnosis in the general population, with a prevalence in the United States of 3-7% in men and 2-5% in women. It is defined as a sleep-related breathing disorder that results in decreased or complete cessation of airflow while the patient has ongoing breathing effort.

It is well documented that trunk position significantly affects the severity of OSA. In fact, 50-75% of individuals with a diagnosis of OSA show supine predominance or worsened apnea-hypopnea index (AHI) when sleeping in the supine position. Positional Obstructive Sleep Apnea (POSA) is defined as an AHI ≥5 with >50% AHI reduction between the supine and non-supine positions and AHI. Studies show 49.5% of individuals with mild OSA (AHI 5-15), 19.4% with moderate OSA (AHI 15-30) and 6.5% in severe OSA (AHI > 30) had POSA. Due to this high prevalence of POSA, especially in the mild and moderate OSA populations, positional therapies have been developed and researched.

In this clinical trial, if only the head position is considered, all subjects are positional sensitive and OSA severity can be calculated and consistently minimized by limiting the allowable range of head roll angle during sleep. Ten subjects underwent a standard polysomnography with an additional head angle sensor and coached to fall asleep in various head positions. Torso position was changed between supine and non-supine for a given head roll angle epoch to show the OSA severity change with torso position. Each sleep epoch of unique head pitch and roll angle was scored individually for AHI and Oxygen Saturation (SPO2) de-saturation.

Investigators hypothesize that specific head roll angles independent of torso position will significantly reduce AHI and SpO2 desaturation severity in patients. The primary aim is to determine the head roll angles that significantly improve POSA independent of torso position. By doing this, Investigators believe to identify a "safe zone" of head roll angles that improve POSA and that can be used to support the development of head positional therapy for POSA patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided written informed consent
* Participant is diagnosed with Positional Obstructive Sleep Apnea
* Participant age is between 21 and 60 years
* If currently on Positive Air Pressure (PAP) therapy, is able to produce compliance data within the last week before screening visit
* Is able to follow directions during the overnight sleep study
* If currently on PAP therapy participant self-report that excessive daytime sleepiness persists when PAP therapy is not in use
* Able to be of "PAP" therapy for 4 nights

Exclusion Criteria:

* Documented diagnosis of Insomnia
* Chronic ear infections
* Persistent neck "pains"
* Persistent chronic posture physical issues
* Previous C-Spine fusion
* History of Cardiac Arrythmia
* History of seizures
* Allergic to Standard Tape used in Sleep Centers
* Non-English speaking.
* Hospitalization within the previous 4 weeks
* Use of antibiotics or steroids within the previous 4 weeks
* Any major uncontrolled disease or condition, such as congestive heart failure, malignancy, end-stage heart disease, end-stage heart disease. Arterial Laterial Sclerosis (ALS), or sever stroke, or other condition as deemed appropriate by investigator as determined by review of medical history and/or participant reported medical history
* History of severe osteoporosis
* Excessive alcohol intake (> 6oz hard liquor, 48 oz beer or 20 oz wine daily), or illicit drug use by review of medical history and/or participant reported medical history
* Daily use of prescribed narcotics (greater than 30 mg morphine equivalent)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-11-19 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacia Sailer, MD, Principal Investigator — Mass Lung and Allergy; Payam Aghazzi, MD, Principal Investigator — Mass Lung and Allergy
Locations (1):
- Mass Lung and Allergy, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual and group subject data for all primary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available immediately after publication. No end date
Access Criteria: Requesters will be required to sign a Data Access Agreement

REFERENCES:
- [Background] Punjabi NM. The epidemiology of adult obstructive sleep apnea. Proc Am Thorac Soc. 2008 Feb 15;5(2):136-43. doi: 10.1513/pats.200709-155MG. PMID 18250205
- [Background] Park JG, Ramar K, Olson EJ. Updates on definition, consequences, and management of obstructive sleep apnea. Mayo Clin Proc. 2011 Jun;86(6):549-54; quiz 554-5. doi: 10.4065/mcp.2010.0810. PMID 21628617
- [Background] Ravesloot MJ, van Maanen JP, Dun L, de Vries N. The undervalued potential of positional therapy in position-dependent snoring and obstructive sleep apnea-a review of the literature. Sleep Breath. 2013 Mar;17(1):39-49. doi: 10.1007/s11325-012-0683-5. Epub 2012 Mar 24. PMID 22441662
- [Background] Epstein LJ, Kristo D, Strollo PJ Jr, Friedman N, Malhotra A, Patil SP, Ramar K, Rogers R, Schwab RJ, Weaver EM, Weinstein MD; Adult Obstructive Sleep Apnea Task Force of the American Academy of Sleep Medicine. Clinical guideline for the evaluation, management and long-term care of obstructive sleep apnea in adults. J Clin Sleep Med. 2009 Jun 15;5(3):263-76. PMID 19960649
- [Background] Mador MJ, Kufel TJ, Magalang UJ, Rajesh SK, Watwe V, Grant BJ. Prevalence of positional sleep apnea in patients undergoing polysomnography. Chest. 2005 Oct;128(4):2130-7. doi: 10.1378/chest.128.4.2130. PMID 16236865
- [Background] Cartwright R, Ristanovic R, Diaz F, Caldarelli D, Alder G. A comparative study of treatments for positional sleep apnea. Sleep. 1991 Dec;14(6):546-52. doi: 10.1093/sleep/14.6.546. PMID 1798889
- [Background] Cartwright RD, Lloyd S, Lilie J, Kravitz H. Sleep position training as treatment for sleep apnea syndrome: a preliminary study. Sleep. 1985;8(2):87-94. doi: 10.1093/sleep/8.2.87. PMID 4012159
- [Background] Jokic R, Klimaszewski A, Crossley M, Sridhar G, Fitzpatrick MF. Positional treatment vs continuous positive airway pressure in patients with positional obstructive sleep apnea syndrome. Chest. 1999 Mar;115(3):771-81. doi: 10.1378/chest.115.3.771. PMID 10084491
- [Background] Permut I, Diaz-Abad M, Chatila W, Crocetti J, Gaughan JP, D'Alonzo GE, Krachman SL. Comparison of positional therapy to CPAP in patients with positional obstructive sleep apnea. J Clin Sleep Med. 2010 Jun 15;6(3):238-43. PMID 20572416
- [Background] Eijsvogel MM, Ubbink R, Dekker J, Oppersma E, de Jongh FH, van der Palen J, Brusse-Keizer MG. Sleep position trainer versus tennis ball technique in positional obstructive sleep apnea syndrome. J Clin Sleep Med. 2015 Jan 15;11(2):139-47. doi: 10.5664/jcsm.4460. PMID 25515276
- [Background] Bignold JJ, Mercer JD, Antic NA, McEvoy RD, Catcheside PG. Accurate position monitoring and improved supine-dependent obstructive sleep apnea with a new position recording and supine avoidance device. J Clin Sleep Med. 2011 Aug 15;7(4):376-83. doi: 10.5664/JCSM.1194. PMID 21897774
- [Background] van Maanen JP, Richard W, Van Kesteren ER, Ravesloot MJ, Laman DM, Hilgevoord AA, de Vries N. Evaluation of a new simple treatment for positional sleep apnoea patients. J Sleep Res. 2012 Jun;21(3):322-9. doi: 10.1111/j.1365-2869.2011.00974.x. Epub 2011 Oct 22. PMID 22017727
- [Background] Levendowski DJ, Seagraves S, Popovic D, Westbrook PR. Assessment of a neck-based treatment and monitoring device for positional obstructive sleep apnea. J Clin Sleep Med. 2014 Aug 15;10(8):863-71. doi: 10.5664/jcsm.3956. PMID 25126032
- [Background] Ravesloot MJL, White D, Heinzer R, Oksenberg A, Pepin JL. Efficacy of the New Generation of Devices for Positional Therapy for Patients With Positional Obstructive Sleep Apnea: A Systematic Review of the Literature and Meta-Analysis. J Clin Sleep Med. 2017 Jun 15;13(6):813-824. doi: 10.5664/jcsm.6622. PMID 28212691
- [Background] van Kesteren ER, van Maanen JP, Hilgevoord AA, Laman DM, de Vries N. Quantitative effects of trunk and head position on the apnea hypopnea index in obstructive sleep apnea. Sleep. 2011 Aug 1;34(8):1075-81. doi: 10.5665/SLEEP.1164. PMID 21804669
- [Background] Gandotra K, May A, Auckley D. Variable Response to CPAP in a Case of Severe Obstructive Sleep Apnea: An Unusual Cause. J Clin Sleep Med. 2018 Jan 15;14(1):145-148. doi: 10.5664/jcsm.6904. PMID 29198296
- [Background] Safiruddin F, Koutsourelakis I, de Vries N. Analysis of the influence of head rotation during drug-induced sleep endoscopy in obstructive sleep apnea. Laryngoscope. 2014 Sep;124(9):2195-9. doi: 10.1002/lary.24598. Epub 2014 Mar 1. PMID 24431007
- [Background] Sleep-related breathing disorders in adults: recommendations for syndrome definition and measurement techniques in clinical research. The Report of an American Academy of Sleep Medicine Task Force. Sleep. 1999 Aug 1;22(5):667-89. No abstract available. PMID 10450601
- [Background] Oksenberg A, Silverberg D, Offenbach D, Arons E. Positional therapy for obstructive sleep apnea patients: A 6-month follow-up study. Laryngoscope. 2006 Nov;116(11):1995-2000. doi: 10.1097/01.mlg.0000237674.66716.a7. PMID 17075418
- See also: Informational website for positional treatment using head pitch and roll angles measuring AHI — http://sleepsystems-llc.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were pre-screened in clinic and using previous sleep study results within a two year time period with a diagnosis of Obstructive Sleep Apnea
Pre-assignment Details: No enrolled participants were excluded
Groups:
- Forehead Sensor Recording Precision Head Pitch and Roll Angle: During an overnight polysomnography, participants were coached by sleep research technologists to sleep with their head in positions hypothesized to minimize apnea severity ≤20⁰ or ≥160⁰, and those hypothesized to maximize apnea severity between 30⁰ and 150⁰. Head roll angles were measured and recorded by the participant's forehead sensor attached with adhesive and tape. Extreme head positions were attempted with the torso in both supine and non-supine positions to show insensitivity to torso position. A custom interface was developed to maintain compatibility with specific bedside polysomnography recorder auxiliary inputs. Sleep epochs were considered those where the subject slept for at least 10 minutes. Each head position epoch was analyzed for apnea hypopnea index and oxygen desaturation. Dual-axis inclinometer attached to the subject's forehead with tape: This is the first clinical trial to address OSA symptom severity and snoring as a direct function of head pitch and roll
Period: Overall Study
Arm/Group | Forehead Sensor Recording Precision Head Pitch and Roll Angle
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 2 participants were disqualified from the study. One participant for no apnea found and one participant found to have central apnea
Groups:
- Forehead Sensor Recording Precision Head Pitch and Roll Angle: During an overnight polysomnography, participants were coached by sleep research technologists to sleep with their head in positions hypothesized to minimize apnea severity ≤20⁰ or ≥160⁰, and those hypothesized to maximize apnea severity between 30⁰ and 150⁰. Head roll angles were measured and recorded by the participant's forehead sensor attached with adhesive and tape. Extreme head positions were attempted with the torso in both supine and non-supine positions so show insensitivity to torso position. A custom interface was developed to maintain compatibility with specific bedside polysomnography recorder auxiliary inputs. Sleep epochs were considered those where the subject slept for at least 10 minutes. Each head position epoch was analyzed for apnea hypopnea index and oxygen desaturation. Dual-axis inclinometer attached to the subject's forehead with tape: This is the first clinical trial to address OSA symptom severity and snoring as a direct function of head pitch and roll.
Arm/Group | Forehead Sensor Recording Precision Head Pitch and Roll Angle
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Apnea Hypopnea Index (AHI) Severity Improvement
Description: Investigators will perform a standard polysomnography with the addition of a precision forehead mounted angular sensor and monitor the severity of apnea hypopnea index (AHI) for the total time duration spent sleeping in each head position. The key measurement is the subjects' relative improvement in AHI with the head supine (45⁰ to 135⁰) as compared to non-supine (<20⁰above the horizon)
Time Frame: 8 hour polysomnography study with subjects being assessed at each head pitch and roll angle epoch
Measure: Count of Participants; unit: Participants
Groups:
- Forehead Sensor Recording Precision Head Pitch and Roll Angle: During an overnight polysomnography, participants were coached by sleep research technologists to sleep with head positions hypothesized to minimize apnea severity ≤20⁰ or ≥160⁰, and those hypothesized to maximize apnea severity between 30⁰ and 150⁰. Head roll angles were measured and recorded by the participant's forehead dual axis inclinometer sensor attached with adhesive and tape. Extreme head positions were attempted with the torso in both supine and non-supine positions so show insensitivity to torso position. Sleep epochs were considered those where the subject slept for at least 10 minutes and each head position epoch was analyzed for apnea hypopnea index and oxygen desaturation. This is the first clinical trial to address Obstructive Sleep Apnea (OSA) symptom severity and snoring as a direct function of head pitch and roll angle. The head pitch and roll angle can be used with high consistency to predict OSA symptom severity.
Arm/Group | Forehead Sensor Recording Precision Head Pitch and Roll Angle
Number analyzed (Participants) | 8
Participants | 8
Statistical Analysis 1: Comparison: Forehead Sensor Recording Precision Head Pitch and Roll Angle; Test type: Other; p < .05, t-test, 2 sided; All statistical tests were completed with a significance of p < 0.05 and 95% confidence intervals. Sample sets were statistically compared and analyzed by using two-tailed, unpaired Student t test analyses of means

2. Primary Outcome: Number of Participants With SpO2 Desaturation Severity Improvement
Description: Investigators will perform a standard polysomnography with the addition of a precision forehead mounted angular sensor and monitor the severity of SpO2 desaturation for the total time duration spent sleeping in each head position. The key measurement is the subjects' relative improvement in SpO2 de-saturation with the head supine (45⁰ to 135⁰) as compared to non-supine (<20⁰above the horizon)
Time Frame: 8 hour polysomnography study with subjects being assessed at each head pitch and roll angle epoch
Measure: Count of Participants; unit: Participants
Arm/Group | Forehead Sensor Recording Precision Head Pitch and Roll Angle
Number analyzed (Participants) | 8
Participants | 8
Statistical Analysis 1: Comparison: Forehead Sensor Recording Precision Head Pitch and Roll Angle; Test type: Other; p < .05, t-test, 2 sided; [other analysis details as in outcome 1, analysis 1]

3. Primary Outcome: Number of Participants With Improvement Independent of Torso Using Forehead Mounted Pitch and Roll Angle Sensor
Description: Investigators will perform a standard polysomnography with the addition of a precision forehead mounted angular sensor and monitor the severity of apnea hypopnea index (AHI) as subjects sleep with the torso in the supine position while the head is ≤ 20⁰ and with the torso in the non-supine position while the head is above 45 degrees. The key measurement is the subjects' relative improvement in AHI with the head supine (45⁰ to 135⁰) as compared to non-supine (<20⁰above the horizon) independent of torso position
Time Frame: 8 hour polysomnography study with subjects being assessed at each head pitch and roll angle epoch
Measure: Count of Participants; unit: Participants
Groups:
- Forehead Sensor Recording Precision Head Pitch and Roll Angle: During an overnight polysomnography, participants were coached by sleep research technologists to sleep with head positions hypothesized to minimize apnea severity ≤20⁰ or ≥160⁰, and those hypothesized to maximize apnea severity between 30⁰ and 150⁰. Head roll angles were measured and recorded by the participant's forehead dual axis inclinometer sensor attached with adhesive and tape. Extreme head positions were attempted with the torso in both supine and non-supine positions so show insensitivity to torso position. Sleep epochs were considered those where the subject slept for at least 10 minutes and each head position epoch was analyzed for apnea hypopnea index and oxygen desaturation. This is the first clinical trial to address OSA symptom severity and snoring as a direct function of head pitch and roll angle. The head pitch and roll angle can be used with high consistency to predict OSA symptom severity.
Arm/Group | Forehead Sensor Recording Precision Head Pitch and Roll Angle
Number analyzed (Participants) | 8
Participants | 8
Statistical Analysis 1: Comparison: Forehead Sensor Recording Precision Head Pitch and Roll Angle; Test type: Other; [other analysis details as in outcome 1, analysis 1]

4. Primary Outcome: Torso Independent With SpO2 Improvement Using Forehead Mounted Pitch and Roll Angle Sensor
Description: Investigators will perform a standard polysomnography with the addition of a precision forehead mounted angular sensor and monitor the severity of SpO2 desaturation as subjects sleep with the torso in the supine position while the head is ≤ 20⁰ and with the torso in the non-supine position while the head is above 45 degrees. The key measurement is the subjects' relative improvement in SpO2 desaturation with the head supine (45⁰ to 135⁰) as compared to non-supine (<20⁰above the horizon) independent of torso position
Time Frame: 8 hour polysomnography study with subjects being assessed at each head pitch and roll angle epoch
Measure: Count of Participants; unit: Participants
Arm/Group | Forehead Sensor Recording Precision Head Pitch and Roll Angle
Number analyzed (Participants) | 8
Participants | 8
Statistical Analysis 1: Comparison: Forehead Sensor Recording Precision Head Pitch and Roll Angle; Test type: Other; p < .05, t-test, 2 sided; [other analysis details as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 8 hours
Description: Serious Adverse Events, All Cause Mortality and Other Adverse Event participants numbers are zero due to the simplistic design of the study. Participants underwent a standard polysomnography with an additional sensor placed on the forehead for data measurements. Participants were monitored and assessed as standard polysomnography testing for any adverse events.
Groups:
- Forehead Sensor Recording Precision Head Pitch and Roll Angle: During polysomnography participants sleep with their head in positions hypothesized to minimize apnea severity ≤20⁰ or ≥160⁰, and those hypothesized to maximize apnea severity between 30⁰ and 150⁰. Head roll angles were measured and recorded by the participant's dual axis accelerometer forehead sensor attached with adhesive and tape. Extreme head positions were attempted with the torso in both supine and non-supine positions so show insensitivity to torso position. Sleep epochs were considered those where the subject slept for at least 10 minutes and each head position epoch was analyzed for apnea hypopnea index and oxygen desaturation. This is the first clinical trial to address OSA symptom severity and snoring as a direct function of head pitch and roll angle. The head pitch and roll angle can be used with high consistency to predict OSA symptom severity. The apnea equation is based on gravitational crush force of the mass of the tongue and nearby tissue on the upper air way.
Arm/Group | Forehead Sensor Recording Precision Head Pitch and Roll Angle
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-04-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT04086407/ICF_000.pdf
  • Study Protocol (2016-04-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT04086407/Prot_001.pdf